CLINICAL TRIAL: NCT02334462
Title: Phase 1 Study of the Safety and Immunogenicity of Pfs230D1M-EPA/Alhydrogel and Pfs25M-EPA/Alhydrogel, a Transmission Blocking Vaccine Against Plasmodium Falciparum Malaria in Adults in the US and Mali
Brief Title: Study of the Safety and Immunogenicity of Pfs230D1M-EPA/Alhydrogel and Pfs25M-EPA/Alhydrogel , a Transmission Blocking Vaccine Against Plasmodium Falciparum Malaria, in Adults in the U.S. and Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Rodolphe Merieux Laboratory@@@Bamako, Mali (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 150044; 15-I-0044
Record Dates: First submitted 2015-01-07; First posted 2015-01-08 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2018-10-22

CONDITIONS: Malaria
Keywords: Assays; Antibody; Reactogenicity; Mosquito; Responses
MeSH Terms: conditions — Malaria | interventions — twinrix; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (7):
- Group 1- Mali (Experimental): Arm A1 (N=5) to receive 16 micrograms Pfs25M on D0, D28 Arm A2 (N=50) to receive 47 micrograms Pfs25M and Normal Saline on D0, D28, D168, D530
  Interventions: Biological: Pfs25M-EPA/Alhydrogel
- Group 1-U.S (Experimental): Arm 1a (N=5) to receive 16 micrograms Pfs25M on D0, D28. Arm 1b (N=5) to receive 47 micrograms Pfs25M on D0, D28.
  Interventions: Biological: Pfs25M-EPA/Alhydrogel
- Group 2- Mali (Experimental): Arm B1 (N=5) to receive 15 micrograms Pfs230D1M on D0, D28 Pfs230D1M-EPA/Alhydrogel Arm B2 (N=50) to receive 40 micrograms Pfs230D1M and Normal Saline on D0, D28, D168, D530
  Interventions: Biological: Pfs230D1M-EPA/Alhydrogel
- Group 2-U.S (Experimental): Arm 2a (N=5) to receive 5 micrograms Pfs230D1M on D0, D28.Arm 2b (N=5) to receive 15 micrograms Pgs230D1M on D0, D28. Arm 2c (N=5) to receive 40 micrograms Pfs230D1M on D0, D28.
  Interventions: Biological: Pfs230D1M-EPA/Alhydrogel
- Group 3- Mali (Experimental): Arm C1 (N=5) to receive 16 micrograms Pfs25M and 15 micrograms Pfs230D1M on D0, D28Arm C2 (N=50) to receive 47 micrograms Pfs25M and 40 microgramsPfs230D1M on D0, D28, D168, D530
  Interventions: Biological: Pfs230D1M-EPA/Alhydrogel; Biological: Pfs25M-EPA/Alhydrogel
- Group 3- U.S. (Experimental): Arm 3a (N=5) to receive 16 micrograms Pfs25M and 15 micrograms Pfs230D1M on D0, D28. Arm 3b (N=5) to receive 47 micrograms Pfs25M and 40 micrograms Pfs230D1M on D0, D28.
  Interventions: Biological: Pfs230D1M-EPA/Alhydrogel; Biological: Pfs25M-EPA/Alhydrogel
- Group 4- Mali (Active Comparator): Arm D1 (N=5) to receive TWINRIX on D0, D28Arm D2 (N=5) to receive TWINRIX and NormalSaline on D0, D28Arm D3 (N=50) to receive TWINRIX and NormalSaline on D0, D28, D168; to receive Menactra andNormal Saline on D530
  Interventions: Drug: TWINRIX; Drug: Menactra

INTERVENTIONS:
Biological: Pfs230D1M-EPA/Alhydrogel
  Arms: Group 2- Mali; Group 2-U.S; Group 3- Mali; Group 3- U.S.
Biological: Pfs25M-EPA/Alhydrogel
  Arms: Group 1- Mali; Group 1-U.S; Group 3- Mali; Group 3- U.S.
Drug: TWINRIX
  Arms: Group 4- Mali
Drug: Menactra
  Arms: Group 4- Mali

SUMMARY:
Background:

- Malaria is a severe infection caused by a parasite. People can get malaria if a mosquito that carries the parasite bites them. Malaria infection does not happen in the United States, but many people in Africa, Asia, and South America are at risk for it. Researchers want to test two vaccines that may help decrease malaria infection.

Objective:

- To see if two vaccines (Pfs25M-EPA/Alhydrogel and Pfs230DIM-EPA/Alhydrogel ) are safe in humans and cause an immune response that will prevent malaria parasites from correctly growing in the mosquito.

Eligibility:

- Healthy adults ages 18 50.

Design:

* There are several groups in this study. Each group will receive a different dose of the vaccine and some groups will received both vaccines.
* Vaccinations will be given on two days about 4 weeks apart.
* Participants will receive each vaccine as an injection into the arm. Blood will be drawn on the day of vaccination.
* In the 4 weeks after receiving a vaccination, participants will have at least 3 clinic visits and 1 phone contact. They will have at least 3 more visits and 3 phone contacts over the next 6 months.
* At each visit, participants will be evaluated for side effects to the vaccine and any new health changes or problems. They will be asked how they are feeling and if they have taken any medicine. Blood and urine samples may be taken at the visit. More follow-up visits may be needed to follow up on changes or problems.

DETAILED DESCRIPTION:
A vaccine to interrupt malaria transmission would be a valuable tool for local elimination or

eradication of this disease. Pfs25 and Pfs230, surface antigens of zygotes and ookinetes in the mosquito stage of Plasmodium falciparum, are the lead candidates for a malaria transmission blocking vaccine. Recombinant Pfs25M and recombinant Pfs230D1M have each been conjugated to Pseudomonas aeruginosa ExoProtein A (EPA) and adjuvanted with Alhydrogel . This dose-escalating phase 1 study will determine safety and immunogenicity of these vaccines in US adults and subsequently in Malian adults.

A total of 260 subjects will be enrolled at sites in the US and Mali to receive escalating doses of Pfs25M- EPA/Alhydrogel , Pfs230D1M-EPA/Alhydrogel , or simultaneous Pfs25MEPA/Alhydrogel and Pfs230D1M-EPA/Alhydrogel . Enrollment within each group will be staggered for additional safety, and subjects will only be enrolled into the simultaneous administration group once each individual dose has been administered and reviewed for safety. Subjects will be followed for at least 6 months after the last vaccination. Safety outcomes will be local and systemic adverse events (AEs) and serious adverse events (SAEs). Immunogenicity outcomes will be antibody responses as measured by ELISA against recombinant Pfs25, Pfs230, and EPA, and B cell responses. Functional activity of the induced antibodies will be assessed by membrane feeding assays conducted at the National Institute of Allergy and Infectious Diseases in the US.

ELIGIBILITY:
* INCLUSION CRITERIA: (US & Mali)

All of the following criteria must be fulfilled for a volunteer to participate in this trial:

1. Age greater than or equal to18 and less than or equal to 50 years.
2. Available for the duration of the trial.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. In good general health and without clinically significant medical history.
5. Females of childbearing potential must be willing to use reliable contraception (as defined below) from 21 days prior to Study Day 0 to 3 months after the last vaccination.

   * Reliable methods of birth control include one of the following: confirmed pharmacologic contraceptives (parenteral) delivery; intrauterine or implantable device.
   * Reliable methods of birth control include concurrent use of a pharmacologic and a barrier method, i.e. two of the following: confirmed pharmacologic contraceptives (oral, transdermal) delivery or vaginal ring AND condoms with spermicide or diaphragm with spermicide.
   * Abstinence of potentially reproductive sexual activity.
   * Non-childbearing women will also be required to report date of last menstrual period, history of surgical sterility (i.e. tubal ligation, hysterectomy) or premature ovarian insufficiency (POI), and will have a baseline urine or serum pregnancy test performed.
6. Willingness to have blood samples stored for future research.
7. Willingness to undergo direct skin feeds (Mali only).
8. Known resident of Bancoumana or surrounding area (Mali only).

EXCLUSION CRITERIA: (US & Mali)

A subject will be excluded from participating in this trial if any one of the following criteria is

fulfilled:

1. Pregnancy as determined by a positive urine or serum human choriogonadotropin ( <=- hCG) test (if female).

   NOTE: Pregnancy is also a criteria for discontinuation of any further dosing or nonsafety related interventions for that subject.
2. Currently breast-feeding (if female).
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol.
4. Hemoglobin, WBC, absolute neutrophils, and platelets outside the local laboratorydefined limits of normal (subjects may be included at the investigator s discretion for not clinically significant values outside of normal range).
5. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal (subjects may be included at the investigator s discretion for not clinically significant values outside of normal range).
6. Infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or

   hepatitis B (HBV).
7. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
8. History of receiving any investigational product within the past 30 days.
9. Participation or planned participation in a clinical trial with an investigational product prior to completion of the follow up visit 28 days following last vaccination OR planned participation in an investigational vaccine study until the last required protocol visit
10. Subject has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
11. History of a severe allergic reaction or anaphylaxis.
12. Severe asthma, defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years.
13. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sj(SqrRoot)(Delta)gren s syndrome, or autoimmune thrombocytopenia.
14. Known immunodeficiency syndrome.
15. Known asplenia or functional asplenia.
16. Use of chronic (greater than or equal to 14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of Study Day 0.
17. Prior to Study Day 0 and every subsequent vaccination day, receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks.
18. Receipt of immunoglobulins and/or blood products within the past 6 months.
19. Previous receipt of an investigational malaria vaccine in the last 5 years.
20. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.
21. Prior malaria infection by history in the last 10 years (US only).
22. Prior travel to a malaria transmission area in the last 5 years or planned travel during the course of the study (US only).
23. History of severe reaction to mosquito bites (Mali only).
24. History of allergy to any component of the comparator vaccine (e.g. neomycin) (Mali only).

    INCLUSION AND EXCLUSION FOR LARGE VOLUME BLOOD DRAW:

    - Individuals previously enrolled in Arms A2, B2, or C2 may be asked to return to the clinic for a single additional visit. This visit would be to collect a single large volume blood sample for additional serological analysis and characterization of B cell receptor usage.

    INCLUSION CRITERIA (LARGE VOLUME BLOOD DRAW):

    -The following criteria must be fulfilled for a volunteer to participate in the large volume blood draw addendum:

    -- Previously enrolled in 15-I-0044 in Arms A2, B2, or C2

    EXCLUSION CRITERIA (LARGE VOLUME BLOOD DRAW):

    - A subject will be excluded from participating in the large volume blood draw addendum if any one of the following criteria is fulfilled:
    * Pregnancy as determined by self report (if female).
    * Within the past 30 days has received a research drug or vaccine or been enrolled in another research drug or vaccine trial.
    * Condition or on a medication that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 538 (Actual)
Dates: Start 2015-01-07; Primary Completion 2016-03-31 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic adverse events and serious advents in U.S. adults and in exposed Malian adults. | U.S. Study: Days 1,3,7,14,28,29,31,35,42,56,84,112,140,168 and 196. Same as U.S. plus Days 169,171,175,182,189,196,203,210,217,240,2 70,300,330,360,390,420,450,480,510,540,541,543,547,554,561,568,575,582,589,610,640,670,700,730

SECONDARY OUTCOMES:
Anti -Pfs25 and Anti-Pfs230 antibody levels elicited by as measured by ELISA in U.S. adults and in exposed Malian adults | U.S. Study: D. 14,28,42,84,140,196 Mali (Safety Arm: Same as the U.S. Mali (Functional Arm): D. 14,28,42,84,140,168,182,196,210,240,300,360,420,480,540,554,568,582,610,670,730

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Farrance CE, Rhee A, Jones RM, Musiychuk K, Shamloul M, Sharma S, Mett V, Chichester JA, Streatfield SJ, Roeffen W, van de Vegte-Bolmer M, Sauerwein RW, Tsuboi T, Muratova OV, Wu Y, Yusibov V. A plant-produced Pfs230 vaccine candidate blocks transmission of Plasmodium falciparum. Clin Vaccine Immunol. 2011 Aug;18(8):1351-7. doi: 10.1128/CVI.05105-11. Epub 2011 Jun 29. PMID 21715576
- [Background] Kaslow DC, Quakyi IA, Syin C, Raum MG, Keister DB, Coligan JE, McCutchan TF, Miller LH. A vaccine candidate from the sexual stage of human malaria that contains EGF-like domains. Nature. 1988 May 5;333(6168):74-6. doi: 10.1038/333074a0. PMID 3283563
- [Background] Shimp RL Jr, Rowe C, Reiter K, Chen B, Nguyen V, Aebig J, Rausch KM, Kumar K, Wu Y, Jin AJ, Jones DS, Narum DL. Development of a Pfs25-EPA malaria transmission blocking vaccine as a chemically conjugated nanoparticle. Vaccine. 2013 Jun 19;31(28):2954-62. doi: 10.1016/j.vaccine.2013.04.034. Epub 2013 Apr 24. PMID 23623858
- [Derived] Cao Y, da Silva Araujo M, Lorang CG, Dos Santos NAC, Tripathi A, Vinetz J, Kumar N. Distinct immunogenicity outcomes of DNA vaccines encoding malaria transmission-blocking vaccine target antigens Pfs230D1M and Pvs230D1. Vaccine. 2025 Feb 15;47:126696. doi: 10.1016/j.vaccine.2024.126696. Epub 2025 Jan 8. PMID 39787798
- [Derived] Sagara I, Healy SA, Assadou MH, Kone M, Swihart BJ, Kwan JL, Fintzi J, Sissoko K, Kamate B, Samake Y, Guindo MA, Doucoure M, Niare K, Dolo A, Diarra B, Rausch KM, Narum DL, Jones DS, MacDonald NJ, Zhu D, Gorres JP, Imeru A, Mohan R, Thera I, Zaidi I, Salazar-Miralles F, Duan J, Neal J, Morrison RD, Muratova O, Sylla D, O'Connell EM, Wu Y, Hume JCC, Coulibaly MB, Anderson CF, Traore SF, Doumbo OK, Duffy PE. Malaria transmission-blocking vaccines Pfs230D1-EPA and Pfs25-EPA in Alhydrogel in healthy Malian adults; a phase 1, randomised, controlled trial. Lancet Infect Dis. 2023 Nov;23(11):1266-1279. doi: 10.1016/S1473-3099(23)00276-1. Epub 2023 Jul 24. PMID 37499679
- [Derived] Fantin RF, Coelho CH, Berhe AD, Magalhaes LMD, Pereira DB, Salinas ND, Tolia NH, Amaratunga C, Suon S, Sagara I, Narum DL, Fujiwara RT, Abejon C, Campos-Neto A, Duffy PE, Bueno LL. Immunological characterization of a VIR protein family member (VIR-14) in Plasmodium vivax-infected subjects from different epidemiological regions in Africa and South America. PLoS Negl Trop Dis. 2023 Apr 7;17(4):e0011229. doi: 10.1371/journal.pntd.0011229. eCollection 2023 Apr. PMID 37027391
- [Derived] Healy SA, Anderson C, Swihart BJ, Mwakingwe A, Gabriel EE, Decederfelt H, Hobbs CV, Rausch KM, Zhu D, Muratova O, Herrera R, Scaria PV, MacDonald NJ, Lambert LE, Zaidi I, Coelho CH, Renn JP, Wu Y, Narum DL, Duffy PE. Pfs230 yields higher malaria transmission-blocking vaccine activity than Pfs25 in humans but not mice. J Clin Invest. 2021 Apr 1;131(7):e146221. doi: 10.1172/JCI146221. PMID 33561016
- [Derived] Guindo A, Sagara I, Ouedraogo B, Sallah K, Assadou MH, Healy S, Duffy P, Doumbo OK, Dicko A, Giorgi R, Gaudart J. "Spatial heterogeneity of environmental risk in randomized prevention trials: consequences and modeling". BMC Med Res Methodol. 2019 Jul 15;19(1):149. doi: 10.1186/s12874-019-0759-z. PMID 31307393